CLINICAL TRIAL: NCT06793124
Title: Comparison of Diagnostic Tests for the Diagnosis of CYTOmegalovirus Organ Disease in Patients With Intestinal BOweL Diseases
Brief Title: Comparison Diagnostic Tests for the Diagnosis of CYTOmegalovirus Organ Disease in Patients With intestinalBOweL Diseases
Acronym: CYTO-BOLD
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: CYTO-BOLD
Record Dates: First submitted 2024-12-01; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Cytomegalovirus (CMV); Inflammatory Bowel Disease (IBD)
Keywords: Cytomegalovirus (CMV); Inflammatory Bowel Disease (IBD); PCR; Tissue biopsy
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * serum samples for CMV-DNA
  * stool samples for CMV-DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with inflammatory bowel disease (IBD): Adult patients with inflammatory bowel disease (IBD) who undergo colonic biopsy for recurrence of the underlying disease

SUMMARY:
Observational, single-center, non-pharmacological, prospective study of adult patients affected by Inflammatory Bowel Disease (IBD) with an ongoing disease exacerbation requiring hospitalization

DETAILED DESCRIPTION:
Patients with chronic inflammatory bowel disease (IBD) are subject to an increased risk of infectious events. This is secondary in part to an intrinsic dysregulation of the immune system, in part to the increasingly frequent need to subject the patient to immunomodulatory therapies for the management of the underlying disease. In this context, it is very difficult from a clinical point of view to be able to demonstrate a concomitant intestinal cytomegalovirus (CMV) organ disease, since the symptoms are often nonspecific or overlapping. Following the guidelines, since there is no well-defined cut-off for viral replication in blood, the gold standard for the diagnosis of intestinal CMV disease remains organ-specific biopsy with immunohistochemical research of the included nuclei. However, at the moment there are no reliable findings for this method that can distinguish a clinically insignificant reactivation from a true organ disease. However, plasma CMV viremia measurement is generally recommended in this setting since active replication in blood could be an epiphenomenon of organ disease. Similarly, some studies have shown a correlation between CMV gastroenteritis and detection of CMV-DNA in fecal samples. Furthermore, several methods have been developed in recent years, and their diagnostic yield has not yet been fully defined. The evaluation of viral load on tissue biopsy by PCR is a method that is gaining ground, and currently the guidelines suggest it in association with immunohistochemistry itself. Some authors suggest a cut-off of 250 cp/mg of tissue to define organ disease. In this setting, the initiation of a specific antiviral treatment remains non-standardized, and it presents expected side effects, primarily bone marrow suppression. However, in several studies, an increased need for surgery for uncontrolled underlying disease has been found in patients with CMV organ disease who are not treated promptly.

From a clinical point of view, in patients who have worsening symptoms related to IBD, being able to identify early markers able to predict CMV colonic organ disease is of crucial importance, since early specific treatment could increase the chances of a favorable outcome, sparing the patient the need for abdominal surgery. In this context, plasma and fecal CMV-DNA dosage represents a rapid diagnostic method, with a turn-over of about 24 hours, which could be an epiphenomenon of the colonic disease itself.

The primary objective of the study is to evaluate the diagnostic performance of different methods used for the diagnosis of CMV infection, namely CMV-DNA on blood and CMV-DNA on fecal samples - comparing them with the gold standard, namely immunohistochemical investigation on biopsy sample in patients affected by IBD with clinical worsening requiring hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years with Inflammatory Bowel Disease (IBD) with worsening of IBD-related symptoms requiring hospital admission
* Signing of informed consent
* Performed endoscopic biopsies to confirm/exclude CMV organ disease

Exclusion Criteria: /

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with inflammatory bowel disease (IBD), either outpatients or requiring hospital admission, who undergo colonic biopsy for recurrence of the underlying disease, will be screened for inclusion
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the diagnostic performance of methods for CMV infection diagnosis | Each samples taken from the patients will be tested through study completion (average of 2 year)
  Evaluation of the diagnostic performance of different methods used for the diagnosis of CMV infection, i.e. CMV-DNA on blood and CMV-DNA on fecal samples - comparing them with the gold standard, i.e. immunohistochemical investigation on biopsy sample in patients affected by IBD with clinical worsening requiring hospitalization

SECONDARY OUTCOMES:
Immunohistochemistry on biopsy sample and PCR for CMV | Each samples taken from the patients will be tested through study completion (average of 2 year)
  Verify the concordance between positive/borderline immunohistochemistry (microscopic examination using specific antibodies to detect the presence of CMV) on biopsy sample and PCR (Polymerase Chain Reaction) for CMV on the sample itself
Immunohistochemical pattern severity and clinical evolution | Each samples taken from the patients will be tested through study completion (average of 2 year)
  Verify if there is a relationship between the severity of the immunohistochemical pattern and clinical evolution and/or the need for major abdominal surgery (colectomy, stoma placement, etc.). Measurement Tools: Immunohistochemistry (Analysis of the severity of the immunohistochemical pattern in biopsy samples, focusing on CMV-related markers); Clinical Assessment (Evaluation of clinical evolution, including the need for major abdominal surgeries)
Evaluation of viral load in biopsy samples | Each samples taken from the patients will be tested through study completion (average of 2 year)
  Verify whether there is a relationship between viral load on biopsy sample and clinical evolution and/or need for major abdominal surgery (colectomy, stoma placement, etc.)
  Correlation between viral load in biopsy samples and clinical outcomes and/or implications for major abdominal surgery (colectomy, stoma placement, etc.)
Evaluation of the Impact of Antiviral Treatment | Each samples taken from the patients will be tested through study completion (average of 2 year)
  Evaluate the impact of an antiviral treatment on clinical evolution and/or need for major abdominal surgery (colectomy, stoma placement, etc.)
Evaluation of clinical evolution of patients with and without CMV organ disease at 30 days | At the follow-up at 30 days (through study completion, an average of 2 year)
  Compare the clinical evolution at 30 days of patients with and without CMV organ disease. The clinical evolution of the patient is understood as the clinical response/refractoriness to medical treatments and the potential need for unplanned major abdominal rescue surgery at the end of the follow-up (+30 days). The clinical response will be evaluated based on the normalization of bowel function (normalization of daily evacuation frequency) and the disappearance of systemic symptoms such as fever, if present, at the end of the follow-up (+30 days).

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Rinaldi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy